CLINICAL TRIAL: NCT01069484
Title: The Effect of Postpartum Pelvic Floor Muscle Training in Women With Injured and Non-injured Pelvic Floor Muscles. A Single Blind Randomized Controlled Trial
Brief Title: Postpartum Pelvic Floor Muscle Training in Women With and Without Injured Pelvic Floor Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: University Hospital, Akershus (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Gunvor Hilde, PT, Msc, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2799004; 2191411 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Incontinence
Keywords: Randomized controlled trial; Post partum pelvic floor muscle training; Urinary incontinence; Pelvic floor dysfunction; Pelvic floor muscle injury; Pelvic floor muscle strength; Pelvic floor muscle morphology
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postpartum pelvic floor muscle training (Experimental): Beyond a customary leaflet (received from the postnatal ward) and the thorough initial instruction on how to contract the PFM correctly, the participants are given supervised pelvic floor muscle group training led by physiotherapists once a week. In addition, the participants train every day at home, with at least 3 sets of 8-12 contractions. Training period is 4 months.
  Interventions: Other: Postpartum pelvic floor muscle training
- Control (No Intervention): Beyond the customary leaflet (received from the postnatal ward) and the thorough initial instruction on how to contract the PFM correctly, the control group participants received no further intervention. They were not discouraged from doing PFMT on their own.

INTERVENTIONS:
Other: Postpartum pelvic floor muscle training — Beyond a customary leaflet and thorough initial instruction on how to contract the PFM correctly, the training participants will attend one weekly supervised exercise class led by an experienced physiotherapist, and perform daily training at home. The intervention starts 6-8 weeks postpartum and last for 4 months. General principles for strength training are followed: 3 sets of 8-12 contractions close to maximum (Bø 1990, Haskell 2007). Emphasis will be on progression in force development. The participants are provided with a DVD of the program (www.corewellness.co.uk). At week 4 during the intervention, the PFM strength will be assessed for each participant. Training adherence at home will be recorded in a training diary, whereas the physical therapist will record group session adherence.
  Other Names: Postpartum PFMT
  Arms: Postpartum pelvic floor muscle training

SUMMARY:
Although pregnancy and childbirth are associated with happiness and a positive life change for most women, it can also be considered as risk periods for injuries to the pelvic floor and development of pelvic floor dysfunction. This may leed to devastating loss of function and quality of life (Ashton-Miller & DeLancey 2007).

The aim of this study is to evaluate the effect of postpartum pelvic floor muscle training for primiparous women with and without pelvic floor muscle injury.

DETAILED DESCRIPTION:
Injuries to the pelvic floor muscles (PFM) and fascias may lead to urinary incontinence (UI), fecal incontinence, pelvic organ prolapse (POP), sensory and emptying abnormalities of the lower urinary tract, defecatory dysfunction, sexual dysfunction and chronic pain syndromes (Bump & Norton 1998, MacLennan et al 2009, Turner et al 2000). Prevalence rates of the most common pelvic floor disorders are generally high in the fertile female population

To date many randomized controlled trials (RCT) have demonstrated significant effect of pelvic floor muscle training (PFMT) in treatment of stress and mixed urinary incontinence, and it is recommended as first line treatment for stress and mixed UI in women (Level I, Grade A) (Abrams 2010). The effect of postpartum PFMT in prevention and treatment of urinary incontinence is investigated in only four RCTs (Sleep 1987, Meyer 2001, Chiarelli 2001, Ewings 2005) and one matched controlled trial (Mørkved 1997). The results are conflicting. The matched controlled trial by Mørkved (1997) shows the far most effective intervention so far, with 50% less prevalence of UI in the training group. Similar results were found for the same long term effect with 50% less prevalence of UI in the training group with the same long term effect (Mørkved 2000). The high effect size may be explained by the close follow-up and relative high training dosage. However, as this was not a RCT, the effect may be overestimated and the trial is often not included in systematic reviews (Hay-Smith 2008).

Only few research groups have measured PFM function and strength, and there are no studies evaluating possible effects of PFMT on PFM injuries and morphology following pregnancy and childbirth. DeLancey (1996) have suggested that the effect of PFMT would be much higher if we knew the causes of incontinence and were able to include only those with intact pelvic floor muscles. This may be true, but the statement also reflects a belief that muscle injury of the PFM cannot be treated with exercise. However, this is in contrast to common practice in treatment of other skeletal muscles e.g. after sport injuries, where all injuries are treated and it is believed that early mobilization and training is important in speeding up tissue healing (Järvinen 2007). Hence, there is a need to conduct a RCT with high methodological and interventional quality (Herbert 2005) to investigate the effect of postpartum PFMT.

ELIGIBILITY:
Inclusion Criteria:

* Primipara women giving birth at Akershus University Hospital, Norway
* Women giving birth to a healthy singleton baby at term
* Women who speak/ understand Scandinavian language

Exclusion Criteria:

* Multiparity
* C-section
* Premature birth (< week 32)
* Prior abortion or stillbirth after 16 weeks of gestation
* Perineal tearing graded as 3b, 3c or 4.
* Illnesses that may interfere with the ability to follow-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, Prof,PhD,PT, Study Director — Norwegian School of Sport Sciences, Dept of Sports Medicine/Akershus University Hospital, Dept of Obstetrics and Gynecology
Locations (1):
- Akershus University Hospital, Dept of Obstetrics and Gynecology, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] Ashton-Miller JA, DeLancey JO. Functional anatomy of the female pelvic floor. Ann N Y Acad Sci. 2007 Apr;1101:266-96. doi: 10.1196/annals.1389.034. Epub 2007 Apr 7. PMID 17416924
- [Background] Bump RC, Norton PA. Epidemiology and natural history of pelvic floor dysfunction. Obstet Gynecol Clin North Am. 1998 Dec;25(4):723-46. doi: 10.1016/s0889-8545(05)70039-5. PMID 9921553
- [Background] Bø K, Hagen RH, Kvarstein B, Jørgensen J, Larsen S. Pelvic floor muscle exercise for the treatment of of female stress urinary incontinence. III. Effects of two different degrees of pelvic floor muscleexercises. Neurourol Urodyn 9:489-502,1990.
- [Background] Bo K, Talseth T, Holme I. Single blind, randomised controlled trial of pelvic floor exercises, electrical stimulation, vaginal cones, and no treatment in management of genuine stress incontinence in women. BMJ. 1999 Feb 20;318(7182):487-93. doi: 10.1136/bmj.318.7182.487. PMID 10024253
- [Background] Chiarelli P, Cockburn J. Promoting urinary continence in women after delivery: randomised controlled trial. BMJ. 2002 May 25;324(7348):1241. doi: 10.1136/bmj.324.7348.1241. PMID 12028976
- [Background] DeLancey JO. Stress urinary incontinence: where are we now, where should we go? Am J Obstet Gynecol. 1996 Aug;175(2):311-9. doi: 10.1016/s0002-9378(96)70140-0. PMID 8765247
- [Background] Ewings P, Spencer S, Marsh H, O'Sullivan M. Obstetric risk factors for urinary incontinence and preventative pelvic floor exercises: cohort study and nested randomized controlled trial. J Obstet Gynaecol. 2005 Aug;25(6):558-64. doi: 10.1080/01443610500231435. PMID 16234140
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Hay-Smith J, Morkved S, Fairbrother KA, Herbison GP. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD007471. doi: 10.1002/14651858.CD007471. PMID 18843750
- [Background] Herbert RD, Bo K. Analysis of quality of interventions in systematic reviews. BMJ. 2005 Sep 3;331(7515):507-9. doi: 10.1136/bmj.331.7515.507. PMID 16141160
- [Background] Jarvinen TA, Jarvinen TL, Kaariainen M, Aarimaa V, Vaittinen S, Kalimo H, Jarvinen M. Muscle injuries: optimising recovery. Best Pract Res Clin Rheumatol. 2007 Apr;21(2):317-31. doi: 10.1016/j.berh.2006.12.004. PMID 17512485
- [Background] MacLennan AH, Taylor AW, Wilson DH, Wilson D. The prevalence of pelvic floor disorders and their relationship to gender, age, parity and mode of delivery. BJOG. 2000 Dec;107(12):1460-70. doi: 10.1111/j.1471-0528.2000.tb11669.x. PMID 11192101
- [Background] Meyer S, Hohlfeld P, Achtari C, De Grandi P. Pelvic floor education after vaginal delivery. Obstet Gynecol. 2001 May;97(5 Pt 1):673-7. doi: 10.1016/s0029-7844(00)01101-7. PMID 11339914
- [Background] Morkved S, Bo K. The effect of postpartum pelvic floor muscle exercise in the prevention and treatment of urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1997;8(4):217-22. doi: 10.1007/BF02765817. PMID 9449300
- [Background] Morkved S, Bo K. Effect of postpartum pelvic floor muscle training in prevention and treatment of urinary incontinence: a one-year follow up. BJOG. 2000 Aug;107(8):1022-8. doi: 10.1111/j.1471-0528.2000.tb10407.x. PMID 10955436
- [Background] Morkved S, Bo K, Schei B, Salvesen KA. Pelvic floor muscle training during pregnancy to prevent urinary incontinence: a single-blind randomized controlled trial. Obstet Gynecol. 2003 Feb;101(2):313-9. doi: 10.1016/s0029-7844(02)02711-4. PMID 12576255
- [Background] Sleep J, Grant A. Pelvic floor exercises in postnatal care. Midwifery. 1987 Dec;3(4):158-64. doi: 10.1016/s0266-6138(87)80035-9. No abstract available. PMID 3320686
- [Background] Turner CE, Young JM, Solomon MJ, Ludlow J, Benness C. Incidence and etiology of pelvic floor dysfunction and mode of delivery: an overview. Dis Colon Rectum. 2009 Jun;52(6):1186-95. doi: 10.1007/DCR.0b013e31819f283f. PMID 19581867
- [Background] Hilde G, Staer-Jensen J, Ellstrom Engh M, Braekken IH, Bo K. Continence and pelvic floor status in nulliparous women at midterm pregnancy. Int Urogynecol J. 2012 Sep;23(9):1257-63. doi: 10.1007/s00192-012-1716-0. Epub 2012 Mar 17. PMID 22426877
- [Background] Hilde G, Staer-Jensen J, Siafarikas F, Gjestland K, Ellstrom Engh M, Bo K. How well can pelvic floor muscles with major defects contract? A cross-sectional comparative study 6 weeks after delivery using transperineal 3D/4D ultrasound and manometer. BJOG. 2013 Oct;120(11):1423-9. doi: 10.1111/1471-0528.12321. Epub 2013 Jul 3. PMID 23834432
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Tennfjord MK, Engh ME, Bo K. The Influence of Early Exercise Postpartum on Pelvic Floor Muscle Function and Prevalence of Pelvic Floor Dysfunction 12 Months Postpartum. Phys Ther. 2020 Aug 31;100(9):1681-1689. doi: 10.1093/ptj/pzaa084. PMID 32367136
- [Derived] Gluppe SL, Hilde G, Tennfjord MK, Engh ME, Bo K. Effect of a Postpartum Training Program on the Prevalence of Diastasis Recti Abdominis in Postpartum Primiparous Women: A Randomized Controlled Trial. Phys Ther. 2018 Apr 1;98(4):260-268. doi: 10.1093/ptj/pzy008. PMID 29351646
- [Derived] Kolberg Tennfjord M, Hilde G, Staer-Jensen J, Siafarikas F, Engh ME, Bo K. Effect of postpartum pelvic floor muscle training on vaginal symptoms and sexual dysfunction-secondary analysis of a randomised trial. BJOG. 2016 Mar;123(4):634-42. doi: 10.1111/1471-0528.13823. Epub 2015 Dec 22. PMID 26691895
- [Derived] Bo K, Hilde G, Staer-Jensen J, Siafarikas F, Tennfjord MK, Engh ME. Postpartum pelvic floor muscle training and pelvic organ prolapse--a randomized trial of primiparous women. Am J Obstet Gynecol. 2015 Jan;212(1):38.e1-7. doi: 10.1016/j.ajog.2014.06.049. Epub 2014 Jun 28. PMID 24983687
- [Derived] Hilde G, Staer-Jensen J, Siafarikas F, Ellstrom Engh M, Bo K. Postpartum pelvic floor muscle training and urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2013 Dec;122(6):1231-8. doi: 10.1097/AOG.0000000000000012. PMID 24201679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant were recruited from a cohort study at Akershus University Hospital (Hilde 2012), or from the hospital's maternity ward or from community health care clinics after giving birth (Hilde 2013).
Groups:
- Postpartum Pelvic Floor Muscle Training: Beyond the customary leaflet (received from the postnatal ward) and the thorough initial instruction on how to contract the pelvic floor muscle (PFM) correctly, the training participants attended a supervised exercise class once a week led by an experienced physiotherapist and were prescribed daily home training over a period of 4 months. The PFM exercise protocol followed general principles for strength training; 3 sets 8-12 contractions close to maximum (Bø et al 1990, Haskell 2007). The participants are provided with a DVD of the program (www.corewellness.co.uk). Training adherence at home was recorded in a training diary whereas the physical therapist recorded group session adherence. Training participants were continuously motivated by the physical therapist to keep up their adherence to training classes and home training, and high performance during training was strongly emphasised.
Period: Overall Study
Arm/Group | Postpartum Pelvic Floor Muscle Training | Control
Started | 87 (27 in the stratum with major levator ani muscle defects and 60 in the stratum without such defects.) | 88 (28 in the stratum with major levator ani muscle defects and 60 in the stratum without such defects.)
Completed | 75 (24 in the stratum with major levator ani muscle defects and 51 in the stratum without such defects.) | 85 (27 in the stratum with major levator ani muscle defects and 58 in the stratum without such defects.)
Not Completed | 12 | 3
Not completed — Death-in-near-family | 1 | 0
Not completed — No specific reason | 8 | 2
Not completed — Illness mother or child | 3 | 1

BASELINE CHARACTERISTICS:
Population: Assuming a similar difference among comparison groups as found by Mørkved and Bø (1997), a two-sided significance of < 0.05 and a power of 0.90 requiered a total of 62 women. For applying stratified analysis on major levator ani (LA) muscle defects, the statistical advice was to aim for 80 women with- and 80 women without major LA muscle defects.
Groups:
- Postpartum Pelvic Floor Muscle Training: Beyond the customary leaflet (received from the postnatal ward) and the thorough initial instruction on how to contract correctly, the training participants attended a supervised exercise class once a week led by an experienced physiotherapist and were prescribed daily home training over a period of 4 months.
- Control: Beyond the customary leaflet (received from the postnatal ward) and the thorough initial instruction on how to contract correctly, the control group received no further intervention.
- Total: Total of all reporting groups
Arm/Group | Postpartum Pelvic Floor Muscle Training | Control | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (4.3) | 30.1 (4.0) | 29.8 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Only primiparous women who delivered a singleton baby vaginally were included. They were included 6 weeks after delivery (mean: 6.1 week, standard deviation: 0.9).
  Participants
    Female | 87 | 88 | 175
    Male | 0 | 0 | 0
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.0 (4.1) | 25.3 (3.9) | 25.7 (4.0)
Level of education [Number; unit: participants]
  College or university | 64 | 79 | 143
  Primary school, high school, other | 23 | 9 | 32
Civil status [Number; unit: participants]
  Married or cohabitant | 80 | 86 | 166
  Single | 7 | 2 | 9
Major defect of the levator ani muscle [Number; unit: participants]
  Major defect | 27 | 28 | 55
  No major defect | 60 | 60 | 120
Urinary Incontinence (Prevalence) [Number; unit: participants]
  Urinary incontinent women | 34 | 44 | 78
  Urinary continent women | 53 | 44 | 97
Urinary incontinence (positive pad test) [Number; unit: participants]
  Positive pad test | 27 | 34 | 61
  Negative pad test | 60 | 54 | 114

OUTCOME MEASURES:

1. Primary Outcome: Urinary Incontinence (Prevalence)
Description: Urinary incontinence was assessed by The International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI Short Form questionnaire, www.iciq.net). Women were considered as incontinent if they reported to leak urine (yes/no) at any frequency.
Time Frame: 6 months postpartum (end of intervention)
Population: Primiparous women who delivered a singleton baby vaginally after more than 32 weeks of gestation. They had to have Scandinavian language skills, no severe perineal tearing, no prior abortion or stillbirth after 16 weeks of gestation, and no illnesses interfering with the ability to follow-up.
Measure: Number; unit: participants
Groups:
- Postpartum Pelvic Floor Muscle Training: Beyond the customary leaflet and the thorough initial instruction on how to contract correctly, the training group attended an exercise intervention for a period of 16 weeks (starting eight 8 weeks after delivery). Once a week the training participants attended a supervised exercise class led by an experienced physical therapist. The exercise class protocol is described in detail by Bø et al (1990) and Mørkved and Bø (1997). Additionally, the training group was prescribed to perform daily pelvic floor muscle training at home (three sets of 8-12 close to maximum contractions).
  Training adherence at home was recorded in a training diary, whereas the physical therapist recorded group session adherence.
Arm/Group | Postpartum Pelvic Floor Muscle Training | Control
Number analyzed (Participants) | 87 | 88
participants
  Urinary incontinent women | 30 | 34
  Urinary continent women | 57 | 54
Statistical Analysis 1: Comparison: Postpartum Pelvic Floor Muscle Training vs Control; Intention to treat was the principal analysis. Missing values for categorical data (self-reported UI) the approach of "last observation carried forward" was used; Test type: Non-Inferiority or Equivalence — Power calculation was based on the study by Mørkved and Bø (1997), showing 67% prevalence reduction of UI in the PFMT group and 34% reduction in the control group. Assuming a similar effect, two-sided significance of <0.05, and a power of 0.90, required a total of 62 women. Stratified analysis on major levator ani (LA) muscle defects was planned, but the effect of PFMT in women with such defects was unknown. The statistical advice was to aim for 80 women with- and 80 women without such defects; p = 0.57, Mantel Haenszel — P-values < 0.05 were considered significant; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.60 to 1.32] — "Pelvic floor muscle training arm" represents the numerator for relative risk and "usual care arm" represents the denominator for relative risk

2. Secondary Outcome: Urinary Incontinence (Positive Pad Test)
Description: Urinary incontinence assessed by pad test, as described by Mørkved and Bø (1997). The cutoff value for a positive test was 2 gram.
  After voiding, the women drank one litre of water. Thirty minutes later they wore a pre-weighted pad and performed a stress test as follows:
  * Jumping up and down with maximal intensity for 30 seconds.
  * Jumping with the legs in alternate abduction and adduction (Jumping Jacks) with maximal intensity for another 30 seconds.
  * Coughing as hard as possible three times. As in the study by Mørkved and Bø (1997), a positive pad-test was set to a cut-off of 2 gram of leakage.
Time Frame: 6 months postpartum (end of intervention)
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Control: Beyond the customary leaflet and the thorough initial instruction on how to contract correctly, the control group received no further intervention..
Arm/Group | Postpartum Pelvic Floor Muscle Training | Control
Number analyzed (Participants) | 87 | 88
participants
  Positive pad test | 19 | 23
  Negative pad test | 68 | 65
Statistical Analysis 1: Comparison: Postpartum Pelvic Floor Muscle Training vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.51, Mantel Haenszel — P-values < 0.05 were considered significant; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.49 to 1.42] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Postpartum Pelvic Floor Muscle Training | Control
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/88
Other Adverse Events (participants affected / at risk) | 0/87 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Postpartum Pelvic Floor Muscle Training (N=87) | Control (N=88)
Any serious adverse effect from pelvic floor muscle training (General disorders) | 0 | 0 — The participants were asked to inform the physiotherapist delivering the intervention if they experienced any serious adverse effect from pelvic floor muscle training. Muscle soreness was not considered as a side effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No